CLINICAL TRIAL: NCT06053086
Title: Adaptive Radiotherapy in Hypersensitive Patients and High Locoregional Risk Breast Cancer With ETHOS Technology
Brief Title: SAHARA-04 : Adaptive Radiotherapy in Hypersensitive Patients and High Locoregional Risk Breast Cancer With ETHOS Technology
Acronym: SAHARA-04
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2023-01 SAH
Record Dates: First submitted 2023-08-23; First posted 2023-09-25 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: radiotherapy; breast cancer; cancer; ETHOS
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: * COHORT A = Treatment ETHOS RT :46 evaluable patients with high risk of LRR and bf+ risk
  * COHORT B = Conventional IMRT : 454 others patients with high risk of LRR and bf- risk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A : Experimental group (Experimental): In cohort A, for patients with high and undetermined risk of fibrosis (bf+), an adaptive BC RT (ETHOS) will be delivered.
  Interventions: Radiation: Treatment ETHOS radiotherapy
- Cohort B : Control group (Active Comparator): In cohort B, for patients with low risk of fibrosis (bf-), an IMRT will be delivered.
  Interventions: Radiation: Conventional IMRT

INTERVENTIONS:
Radiation: Treatment ETHOS radiotherapy — • Cohort A: Adaptive RT: PTV = CTV + 2 mm (except for IMC with 5mm), excluding 5mm beneath the skin
  Arms: Cohort A : Experimental group
Radiation: Conventional IMRT — • Cohort B: IMRT: PTV = CTV + 7mm, excluding 5mm beneath the skin
  Arms: Cohort B : Control group

SUMMARY:
* Prospective, open-label, bi-center study, assessing the clinical outcomes of adaptive breast radiotherapy with ETHOS in hypersensitive patients.
* Bi-centric with ETHOS center : ICM (Institut du Cancer de Montpellier) and ISC (Institut Sainte Catherine) Avignon
* 500 patients will be included:
* COHORTE A = Treatment ETHOS RT :46 evaluable patients with high risk of LRR and bf+ risk
* COHORT B = Conventional IMRT : 454 others patients with high risk of LRR and bf- risk

DETAILED DESCRIPTION:
1. Breast cancer (BC) patients with high risk of severe radio-induced side effects

   Severe but also moderate toxicities after curative-intent radiotherapy (RT), such as fibrosis, retraction or telangiectasia can have a negative impact on quality of life and a marked effect on subsequent psychological outcome. A number of factors are known to increase the risk of radiation toxicity including individual radiosensitivity. While toxicity risks for populations of patients are known, the determination of an individual's normal tissue radiosensitivity is seldom possible before treatment.

   Therefore, current practice standards commonly prescribe radiation dose according to clinical scenarios, without regard to the genotype or phenotype of the individual being irradiated.

   In that context, several teams have developed and validated prospectively or retrospectively (a rapid (72 h) radiosensitivity assay based on flow cytometric assessment of radiation-induced CD8 T-lymphocyte apoptosis (RILA).

   An excellent negative predictive value was found in the case of high RILA value and grade 0-1 late toxicity in breast cancers.

   In addition, all severe side-effects (grade ≥2) were observed in patients with low values of RILA.

   Recently, the REQUITE consortium aimed to establish a resource for multi-national validation of models and biomarkers that predict risk of late toxicity following radiotherapy.

   This international, prospective cohort study recruited cancer patients in 26 hospitals in eight countries between April 2014 and March 2017.

   RILA assay data were available for 1319 patients. More recently, at the last ESTRO Annual Meeting in Milan (April 2019), this Consortium found that low RILA was associated with long-term side effects such breast fibrosis (bf+) after adjuvant BC radiotherapy.

   The median value of RILA was 9.51% in patients with grade ≥2 bf+ (n=17) vs. 17.15% in patients without toxicity (n=631), p=0.003. In the meantime, the German team presented results from a large prospective ISE cohort with a very long-term follow-up (median FU=11.6 years). High RILA values were inversely correlated with the risk of fibrosis (p=0,011) and telangiectasia (p<0.001). Univariate ROC analysis and multivariate analysis showed higher AUC and c-stat values outside than within the surgical area.

   With a level one of clinical evidence, the RILA assay is recommended by the French guidelines since 2022. The RILA assay has now clear potential to be a useful biomarker for selecting individuals likely to display an increased probability of toxicity to RT. A French Company (NovaGray) now industrializes this assay (NovaGray RILA Breast®).
2. BC patients with high risk of locoregional relapse (LRR)

   Node positive (pN+) patients after breast conserving surgery (BCS) and adjuvant systemic therapies had a high risk of LRR (among 16%) with most of LRR which occurred within 5 years.

   Significant improvements of distant free survival (DFS) were observed in case of regional nodes irradiation in large phase III trials: the EORTC 22922/10925 trial and the MA20 trial. In addition, adjuvant postmastectomy radiotherapy (PMRT) is a standard of care after radical mastectomy in case of nodal involvement as chest wall and regional nodes irradiation reduced both recurrence and breast cancer mortality in particular in BC patients with one to three positive lymph nodes even when systemic therapy was given.

   Therefore, there is a need in those pN+ BC patient's population to well cover planning target volume (PTV) of whole breast (WB) or chest wall (CW) and regional nodes. Intensity-modulated radiotherapy (IMRT) is an appropriate technique to that end.
3. Personalized radiotherapy in BC patients with high risk of LRR and bf+ risk

The present study aimed to assess acute and late toxicities after adaptive radiotherapy ETHOS in high risk of LRR and hypersensitive breast cancer (bf+ BC) patients.

The investigators propose, in high risk of LRR/ bf+ BC patients, to reduce PTVs thanks to ETHOS technology, an adaptive image-guided IMRT radiotherapy.

Usually, PTVs are generated by adding 7 mm-margins around CTVs. By decreasing intrafraction variability, PTV margins could be significantly reduced closed to clinical target volume (CTV). Therefore, target volumes will be significantly reduced.

In an adaptive radiotherapy a new plan is generated every fraction based on the organ and clinical target volume (CTV) delineations of that fraction. With these daily adaptations, inter fractions modifications are taken into account.

The hypothesis is therefore that acute and late RT side effects occurring after ETHOS adaptive RT in bf+ BC patients will not be superior than those obtained after IMRT RT in BC non-hypersensitive patients.

This hypothesis is based on a personalized approach (driven by a predictive assay of late effects to select patients with high and undetermined risk toxicity: for each patient, NovaGray will provide a report including the result of the NovaGray RILA Breast® test as well as a binary risk category (low risk or undetermined risk or high risk).

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old.
* Conservative breast cancer surgery or radical mastectomy.
* At least pN1 breast cancers, regardless breast cancer subtypes.
* Tumor negative margins.
* Indication of whole breast and node irradiation.
* Extension evaluation of disease will be proven negative (M0).
* Risk level of breast fibrosis identified by the centralized NovaGray RILA Breast® test
* Must be geographically accessible for follow-up.
* Written and dated informed consent.
* Affiliated to the French national social security system.

Exclusion Criteria:

* Patients with distant metastases.
* Bilateral breast cancer (concomitant or prior) except in situ lesion, either ductal or lobular, of the contralateral breast.
* Patients with previous or concomitant other (not breast cancer) malignancy within the past 5 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who have had a previous other malignancy must have been disease free for at least five years.
* Patients with other non-malignant systemic diseases (cardiovascular, renal, hepatic, lung embolism, etc.) which would prevent prolonged follow-up.
* Patients treated with systemic investigational drugs within the past 30 days (Observational cohorts are accepted if the collection of data does not interfere with the current trial)
* Untreated hypothyroidism
* Patients known to be HIV positive (no specific tests are required to determine the eligibility).
* Patients known as hypersensitive to radiation (ATM Homozygote, p53-/-,…)
* Pregnant or breast-feeding women
* Patient unable to comply with study obligations for geographic, social, or physical reasons, or who is unable to understand the purpose and procedures of the study
* Person deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer
Enrollment: 500 (Estimated)
Dates: Start 2025-03-06 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Rate of patients without any grade 2 and more toxicities within the planning target volume | at 3 years
  A toxicity of grade 2 and more is defined as an observation of grade 2 and more, in case of late toxicities it should be at least confirmed by two consecutive visits.

SECONDARY OUTCOMES:
rate of Acute & late toxicity | From the start of RT to 12 weeks post RT and from 12 weeks post RT to 3 years post RT
  acute toxicity is defined as side effects observed from the start of RT to 12 weeks post RT, according to NCI-CTCAE v5. Late toxicity is defined as side effects observed from 12 weeks post RT to 3 years post RT, according to NCI-CTCAE v5
Quality of life by using QLQ-C30 (and BR 23 module) questionnaire score | at 0/3/6/12/18/24/30/36 months post RT
  score obtained by assessed questionnaires
Quality of life by using GPAQ questionnaire score | at 0/3/6/12/18/24/30/36 months post RT
  score obtained by assessed questionnaires
Quality of life by using MFI questionnaire score | at 0/3/6/12/18/24/30/36 months post RT
  score obtained by assessed questionnaires
Local recurrence rate (LRR) | at 3 years
  LRR will be deducted from the local recurrence survival defined as the interval between date of inclusion and the occurrence of local relapse. Patients without relapse at the analysis will be censored at the date of last follow-up
Relapse-free survival (RFS) rate | at 3 years
  RFS is defined as the interval between date of inclusion and the occurrence of relapse. Patients without relapse at the analysis will be censored at the date of last follow-up
Time to severe RT toxicities rate | at 3 years
  Time to severe RT toxicities is defined as the interval between date of inclusion and the occurrence of radio-induced Gr2+ toxicities (i.e. event). Patients without event at the analysis will be censored at the date of last follow-up.
Overall survival (OS) rate | at 3 years
  OS is defined as the interval between date of inclusion and the occurrence of death, due to any cause. Patients alive at the analysis will be censored at the date of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: BOURGIER CELINE, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle; ARNAUD ANTOINE, Principal Investigator — INSTITUT SAINTE CATHERINE / AVIGNON
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No